CLINICAL TRIAL: NCT02633501
Title: P03277 Dose Finding Study in Central Nervous System (CNS) Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GDX-44-004
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: CNS Lesion; Blood Brain Barrier Defect
MeSH Terms: interventions — gadopiclenol; gadobenic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subset 1 Arm 1 (Experimental): One of the two doses of P03277 (0.05 or 0.1 mmol/kg)-enhanced MRI then gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
  Interventions: Drug: P03277; Drug: Gadobenate dimeglumine; Device: MRI
- Subset 1 Arm 2 (Experimental): Gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI then one of the two doses of P03277 (0.05 or 0.1 mmol/kg)-enhanced MRI
  Interventions: Drug: P03277; Drug: Gadobenate dimeglumine; Device: MRI
- Subset 2 Arm 1 (Experimental): One of the four doses of P03277 (0.025, 0.05, 0.1 or 0.2 mmol/kg)-enhanced MRI then gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
  Interventions: Drug: P03277; Drug: Gadobenate dimeglumine; Device: MRI
- Subset 2 Arm 2 (Experimental): Gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI then one of the four doses of P03277 (0.025, 0.05, 0.1 or 0.2 mmol/kg)-enhanced MRI
  Interventions: Drug: P03277; Drug: Gadobenate dimeglumine; Device: MRI

INTERVENTIONS:
Drug: P03277 — Single intravenous (IV) bolus injection at a rate of 2 mL/second
  Other Names: Gadopiclenol
Drug: Gadobenate dimeglumine — Single IV bolus injection at a rate of 2 mL/second
  Other Names: MultiHance
Device: MRI

SUMMARY:
The purpose of this study was to determine a safe and effective dose of a new gadolinium-based contrast agent (GBCA) P03277 based on the Contrast to Noise Ratio (CNR) when comparing with gadobenate dimeglumine (MultiHance®) at 0.1 mmol/kg body weight (BW).

Contrast to Noise Ratio (CNR), a well-known quantitative parameter directly related to contrast medium/GBCA efficacy, was chosen as the primary endpoint in order to have a precise determination of P03277 clinical dose.

This was a multi-center, international, prospective, double-blind, randomized, controlled, parallel dose groups, cross-over with comparator study in male and female subjects presenting with known or highly suspected focal areas of disruption of the Blood Brain Barrier including at least one expected enhancing lesion of minimum 5 mm, who were scheduled to undergo a routine contrast-enhanced Magnetic Resonance Imaging (MRI) of Central Nervous System.

DETAILED DESCRIPTION:
Two subsets of subjects were included in the study:

* The subset 1 included the first randomized subject of each study center. Subjects were randomly assigned in a 1:1 ratio to receive 0.05 or 0.1 mmol/kg BW of P03277 and 0.1 mmol/kg BW of gadobenate dimeglumine.
* Subset 2 was composed of all subjects (except the first one of each study center) selected by the study center. Subjects were randomly assigned in a 1:1:1:1 ratio to receive 0.025, 0.05, 0.1 or 0.2 mmol/kg BW of P03277 and 0.1 mmol/kg BW of gadobenate dimeglumine.

During the course of the study, two MRIs were obtained from each subject: one unenhanced and P03277-enhanced MRI; and one unenhanced and gadobenate dimeglumine-enhanced MRI. MRI images were evaluated off-site by 3 independent blinded readers for the primary endpoint (CNR).

ELIGIBILITY:
Inclusion Criteria:

* Female or male adult subjects, with known or highly suspected focal areas of disrupted Blood Brain Barrier including at least one expected enhancing lesion of minimum 5 mm (long axis). This lesion had been detected on a previous imaging procedure (computerized Tomography [CT] or MRI).
* Subject scheduled for a routine contrast-enhanced MRI examination of Central Nervous System for clinical reasons and agreeing to have a second contrast-enhanced MRI examination for the purpose of the study.

Exclusion Criteria:

* Subject presenting with acute or chronic Grade III (at least) renal insufficiency, defined as an estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m² based on one eGFR assessment performed the day of the MRI prior to the first contrast agent injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin BENDSZUS, MD, Principal Investigator — University Hospital Heidelberg
Locations (28):
- United States (10):
  - Northwestern memorial hospital, Chicago, Illinois
  - Beth israel deaconess medical center, Boston, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Penn State milton S. Hershey Medical center, Hershey, Pennsylvania
  - University of Pensylvania medical center, Philadelphia, Pennsylvania
  - Temple university hospital, Philadelphia, Pennsylvania
  - Rhode Island hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of texas McGovern medical school, Houston, Texas
  - University of Washington, Seattle, Washington
- Belgium (2):
  - ZNA campus Middelheim, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
- Fakultni nemocnice Olomouc, Olomouc, Czechia
- Hungary (2):
  - Neurology Clinic-Semmelweis Medical University, Budapest
  - Pecsi Tudomany Egyetem Klinikai kozpont Idegsebeszeti Klinica, Pécs
- Italy (4):
  - Ospedali Riuniti di Ancona, Ancona
  - Ospedale san Raffaele, Milan
  - AO S. Andrea Universita La Sapienza, Roma
  - Azienda policlinico Umberto, Roma
- Mexico (3):
  - Centro medico ABC santa fe, Mexico City
  - Axis heilsa, Monterrey
  - Clinical research institute SC, Tlalnepantla
- Poland (3):
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Oddzial w Gliwicach, Gliwice
  - krakowski Szpital specjalistyczny il Jana Pawla II, Krakow
  - Samodzielny publiczny szpital, Lublin
- South Korea (3):
  - Asan medical center, Seoul
  - Samsung medical center, Seoul
  - Seoul National university hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 312 screened subjects, 32 subjects were screening failure. 280 subjects were randomized: 28 in subset 1 and 252 in subset 2. Images from the subset 1 were used for training of off-site readers and validation of imaging protocol. Consequently, these subjects were not included in the efficacy analysis but only in the safety assessment.
Groups:
- Subset 1 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine; Subset 2 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine: P03277 (0.05 mmol/kg)-enhanced MRI then gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI or vice versa
  P03277: Single intravenous (IV) bolus injection at a rate of 2 mL/second
  Gadobenate dimeglumine: Single IV bolus injection at a rate of 2 mL/second
- Subset 1 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine; Subset 2 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine: P03277 (0.1 mmol/kg)-enhanced MRI then gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI or vice versa
  P03277: Single intravenous (IV) bolus injection at a rate of 2 mL/second
  Gadobenate dimeglumine: Single IV bolus injection at a rate of 2 mL/second
- Subset 2 - P03277 0.025 mmol/kg/Gadobenate Dimeglumine: P03277 (0.025 mmol/kg)-enhanced MRI then gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI or vice versa
  P03277: Single intravenous (IV) bolus injection at a rate of 2 mL/second
  Gadobenate dimeglumine: Single IV bolus injection at a rate of 2 mL/second
- Subset 2 - P03277 0.2 mmol/kg/Gadobenate Dimeglumine: P03277 (0.2 mmol/kg)-enhanced MRI then gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI or vice versa
  P03277: Single intravenous (IV) bolus injection at a rate of 2 mL/second
  Gadobenate dimeglumine: Single IV bolus injection at a rate of 2 mL/second
Period: Overall Study
Arm/Group | Subset 1 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine | Subset 1 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine | Subset 2 - P03277 0.025 mmol/kg/Gadobenate Dimeglumine | Subset 2 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine | Subset 2 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine | Subset 2 - P03277 0.2 mmol/kg/Gadobenate Dimeglumine
Started | 14 | 14 | 62 | 63 | 64 | 63
Completed | 12 | 11 | 55 | 59 | 53 | 48
Not Completed | 2 | 3 | 7 | 4 | 11 | 15
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 2 | 1 | 3
Not completed — Various other reasons | 0 | 2 | 4 | 1 | 7 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Subjects of subset 1 were only included in the safety assessment. The Full Analysis Set included 240 subjects from subset 2 who had available results for CNR from both unenhanced and enhanced measurements derivable from one MRI by at least one off-site reader. Analyses using the FAS were based on the contrast agent allocated by the randomization.
Groups:
- Subset 2 - P03277 0.025 mmol/kg/Gadobenate Dimeglumine: P03277 (0.025 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
- Subset 2 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine; Subset 1 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine: P03277 (0.05 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
- Subset 2 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine; Subset 1 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine: P03277 (0.1 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
- Subset 2 - P03277 0.2 mmol/kg/Gadobenate Dimeglumine: P03277 (0.2 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
- Total: Total of all reporting groups
Arm/Group | Subset 2 - P03277 0.025 mmol/kg/Gadobenate Dimeglumine | Subset 2 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine | Subset 2 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine | Subset 2 - P03277 0.2 mmol/kg/Gadobenate Dimeglumine | Subset 1 - P03277 0.05 mmol/kg/Gadobenate Dimeglumine | Subset 1 - P03277 0.1 mmol/kg/Gadobenate Dimeglumine | Total
Number analyzed (Participants) | 57 | 62 | 61 | 60 | 14 | 14 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.9) | 54.0 (14.8) | 54.2 (14.4) | 52.1 (13.7) | 54.9 (13.3) | 56.1 (16) | 53.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 30 | 39 | 10 | 5 | 157
  Male | 23 | 23 | 31 | 21 | 4 | 9 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 8 | 5 | 8 | 4 | 2 | 1 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 4 | 2 | 2 | 2 | 12
  White | 47 | 55 | 49 | 54 | 10 | 11 | 226
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Contrast to Noise Ratio (CNR) Difference
Description: The Contrast-to-Noise Ratio (CNR) was calculated from the signal intensity measurement of maximum 3 enhanced lesions by 3 independent blinded readers. Only lesions detected by both MRIs after lesion tracking were used. The difference in CNR was calculated as follow: CNR (P03277) - CNR (gadobenate dimeglumine).
Time Frame: 1 day procedure
Population: The analysis was done for each of the 3 independent off-site readers using the Per Protocol Set that included all subjects without major protocol deviations. A subject was analyzed as soon as he had a matching evaluation of the CNR at both MRIs by at least 1 off-site reader. Therefore, the numbers of subjects analyzed by reader could be different.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Groups:
- P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 1; P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 2; P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 3: P03277 (0.025 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
- P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 1; P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 2; P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 3: P03277 (0.05 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
- P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 1; P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 2; P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 3: P03277 (0.1 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
- P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 1; P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 2; P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 3: P03277 (0.2 mmol/kg)-enhanced MRI and gadobenate dimeglumine (0.1 mmol/kg)-enhanced MRI
Arm/Group | P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 1 | P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 1 | P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 1 | P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 1 | P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 2 | P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 2 | P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 2 | P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 2 | P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 3 | P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 3 | P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 3 | P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 3
Number analyzed (Participants) | 54 | 56 | 51 | 44 | 44 | 47 | 43 | 41 | 49 | 51 | 45 | 42
Ratio | -10.59 [-14.59 to -6.58] | 2.18 [-2.67 to 7.03] | 8.66 [3.52 to 13.79] | 14.45 [7.64 to 21.25] | -14.14 [-23.33 to -4.95] | 1.91 [-7.28 to 11.10] | 19.38 [11.42 to 27.34] | 38.37 [18.62 to 58.12] | -23.96 [-33.78 to -14.13] | 2.47 [-8.39 to 13.32] | 29.23 [16.05 to 42.41] | 51.96 [30.36 to 73.55]
Statistical Analysis 1: Comparison: P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 1; Holm's Step-Down Method; Test type: Superiority; Mixed Models Analysis — Testing procedure stopped; Least Squares Mean = -10.59, Standard Error of Mean 2.00
Statistical Analysis 2: Comparison: P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 1; Holm's Step-Down Method; Test type: Superiority; p = 0.1858, Mixed Models Analysis — Superiority not confirmed; Least Squares Mean = 2.18, Standard Error of Mean 2.42
Statistical Analysis 3: Comparison: P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 1; Holm's Step-Down Method; Test type: Superiority; p = 0.0007, Mixed Models Analysis — Superiority confirmed; Least Squares Mean = 8.66, Standard Error of Mean 2.55
Statistical Analysis 4: Comparison: P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 1; Holm's Step-Down Method; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Superiority confirmed; Least Squares Mean = 14.45, Standard Error of Mean 3.37
Statistical Analysis 5: Comparison: P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 2; Holm's Step-Down Method; Test type: Superiority; Mixed Models Analysis — Testing procedure stopped; Least Squares Mean = -14.14, Standard Error of Mean 4.55
Statistical Analysis 6: Comparison: P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 2; Holm's Step-Down Method; Test type: Superiority; p = 0.3384, Mixed Models Analysis — Superiority not confirmed; Least Squares Mean = 1.91, Standard Error of Mean 4.56
Statistical Analysis 7: Comparison: P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 2; Holm's Step-Down Method; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Superiority confirmed; Least Squares Mean = 19.38, Standard Error of Mean 3.94
Statistical Analysis 8: Comparison: P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 2; Holm's Step-Down Method; Test type: Superiority; p = 0.0002, Mixed Models Analysis — Superiority confirmed; Least Squares Mean = 38.37, Standard Error of Mean 9.76
Statistical Analysis 9: Comparison: P03277 0.025 mmol/kg - Gadobenate Dimeglumine - Reader 3; Holm's Step-Down Method; Test type: Superiority; Mixed Models Analysis — Testing procedure stopped; Least Squares Mean = -23.96, Standard Error of Mean 4.88
Statistical Analysis 10: Comparison: P03277 0.05 mmol/kg - Gadobenate Dimeglumine - Reader 3; Holm's Step-Down Method; Test type: Superiority; p = 0.3249, Mixed Models Analysis — Superiority not confirmed; Least Squares Mean = 2.47, Standard Error of Mean 5.4
Statistical Analysis 11: Comparison: P03277 0.1 mmol/kg - Gadobenate Dimeglumine - Reader 3; Holm's Step-Down Method; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Superiority confirmed; Least Squares Mean = 29.23, Standard Error of Mean 6.53
Statistical Analysis 12: Comparison: P03277 0.2 mmol/kg - Gadobenate Dimeglumine - Reader 3; Holm's Step-Down Method; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Superiority confirmed; Least Squares Mean = 51.96, Standard Error of Mean 10.68

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from informed consent signature up to one day after the second MRI, up to 22 days
Description: The Safety Set included all subjects (from both subsets 1 and 2) who had received at least one injection of contrast agent, regardless of the quantity.
Groups:
- P03277 0.025 mmol/kg: Patients who received one injection of P03277 0.025 mmol/kg regardless of injection order vs gadobenate dimeglumine (subset 2).
- P03277 0.05 mmol/kg: Patients who received one injection of P03277 0.05 mmol/kg regardless of injection order vs gadobenate dimeglumine (subset 1 + subset 2).
- P03277 0.1 mmol/kg: Patients who received one injection of P03277 0.1 mmol/kg regardless of injection order vs gadobenate dimeglumine (subset 1 + subset 2)
- P03277 0.2 mmol/kg: Patients who received one injection of P03277 0.2 mmol/kg regardless of injection order vs gadobenate dimeglumine (subset 2)
- Gadobenate Dimeglumine: Patients who received one injection of gadobenate dimeglumine regardless of injection order vs P03277 (subset 1 + subset 2).
Arm/Group | P03277 0.025 mmol/kg | P03277 0.05 mmol/kg | P03277 0.1 mmol/kg | P03277 0.2 mmol/kg | Gadobenate Dimeglumine
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/74 | 0/70 | 0/56 | 0/256
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/74 | 1/70 | 1/56 | 2/256
Other Adverse Events (participants affected / at risk) | 14/56 | 12/74 | 19/70 | 18/56 | 57/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P03277 0.025 mmol/kg (N=56) | P03277 0.05 mmol/kg (N=74) | P03277 0.1 mmol/kg (N=70) | P03277 0.2 mmol/kg (N=56) | Gadobenate Dimeglumine (N=256)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningioma surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — After injection of P03277 at 0.1 mmol/kg.
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — After injection of P03277 at 0.2 mmol/kg
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | P03277 0.025 mmol/kg (N=56) | P03277 0.05 mmol/kg (N=74) | P03277 0.1 mmol/kg (N=70) | P03277 0.2 mmol/kg (N=56) | Gadobenate Dimeglumine (N=256)
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 2
Peripheral coldness (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 2 | 5 | 7 | 9
Injection site coldness (General disorders) | 1 | 0 | 1 | 0 | 4
Fatigue (General disorders) | 2 | 0 | 0 | 2 | 1
Injection site warmth (General disorders) | 0 | 1 | 0 | 0 | 3
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 2
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 2
Injection site oedema (General disorders) | 1 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1
Injection site bruising (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 2 | 0
Injection site inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Blood pressure increased (Investigations) | 2 | 0 | 1 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 2
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT interval abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 0 | 0
Urobilinogen urine (Investigations) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 3 | 1 | 0 | 7
Diziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 4
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 9
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 2 | 1 | 1 | 5
Bilirubinuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 4
Glycosuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 3
Haemoglobinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 5
Proteinuria (Renal and urinary disorders) | 1 | 2 | 1 | 1 | 2
Ketonuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Nitrituria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 1 | 4
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 — No post-injection adverse events occurred
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 — No post-injection adverse events occurred
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 — No post-injection adverse events occurred
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 — No post-injection adverse events occurred
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 1 — No post-injection adverse events occurred
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 — No post-injection adverse events occurred
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 — No post-injection adverse events occurred
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 — No post-injection adverse events occurred
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 — No post-injection adverse events occurred
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 — No post-injection adverse events occurred
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 — No post-injection adverse events occurred

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT02633501/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02633501/SAP_003.pdf